CLINICAL TRIAL: NCT03560752
Title: CMV-MVA Triplex Vaccination of Stem Cell Donors to Enhance CMV Specific Immunity and Prevent CMV Viremia in Recipients After Stem Cell Transplant
Brief Title: CMV-MVA Triplex Vaccination of Stem Cell Donors in Preventing CMV Viremia in Participants With Allogeneic Transplant
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18007; NCI-2018-01115 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18007 (Other: City of Hope Medical Center)
Record Dates: First submitted 2018-06-07; First posted 2018-06-18 (Actual); Results first posted 2024-01-31 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Accelerated Phase CML, BCR-ABL1 Positive; Acute Lymphoblastic Leukemia in Remission; Acute Myeloid Leukemia in Remission; Chronic Lymphocytic Leukemia; Chronic Phase CML, BCR-ABL1 Positive; Cytomegalovirus Positive; Donor; Hematopoietic Cell Transplant Recipient; Hodgkin Lymphoma; Myelodysplastic Syndrome; Myelodysplastic/Myeloproliferative Neoplasm; Non-Hodgkin Lymphoma; Myelofibrosis; Hematopoietic and Lymphoid Cell Neoplasm
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Chronic-Phase; Hodgkin Disease; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Lymphoma, Non-Hodgkin; Primary Myelofibrosis; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Donor (multi-peptide CMV-modified vaccinia Ankara vaccine) (Experimental): Donors receive multi-peptide CMV-modified vaccinia Ankara vaccine injection between days -60 and -10 prior to granulocyte colony stimulating factor mobilization.
  Interventions: Biological: Multi-peptide CMV-Modified Vaccinia Ankara Vaccine
- Receipient (multi-peptide CMV-modified vaccinia Ankara vaccine) (Experimental): Participants undergo hematopoietic cell transplantation on day 0 and receive multi-peptide CMV-modified Vaccinia Ankara vaccine injection on days 28 and 56.
  Interventions: Biological: Multi-peptide CMV-Modified Vaccinia Ankara Vaccine

INTERVENTIONS:
Biological: Multi-peptide CMV-Modified Vaccinia Ankara Vaccine — Given via injection
  Other Names: CMV-MVA Triplex Vaccine

SUMMARY:
This phase II trial studies how well multi-peptide CMV-modified vaccinia Ankara (CMV-MVA Triplex) vaccination of stem cell donors works in preventing cytomegalovirus (CMV) viremia in participants with blood cancer undergoing donor stem cell transplant. Giving a vaccine to the donors may boost the recipient's immunity to this virus and reduce the chance of CMV disease after transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish the feasibility and safety of priming CMV immunity in donors by Triplex vaccination prior to peripheral blood stem cell (PBSC) harvest.

SECONDARY OBJECTIVES:

I. Examine if Triplex vaccination of hematopoietic stem cell transplant (HCT) donors has an impact on CMV events.

OUTLINE:

Donors receive multi-peptide CMV-modified vaccinia Ankara vaccine injection between days -60 and -10 prior to granulocyte colony stimulating factor mobilization. Participants undergo hematopoietic cell transplantation on day 0.

After completion of study treatment, participants are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* DONOR: Ability to comprehend the investigational nature of the study and provide informed consent
* DONOR: Willing to receive Triplex vaccination, a minimum of 14 days prior to the PBSC collection
* DONOR VACCINATION: Donors are eligible to be vaccinated prior to the determination of their human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV) and human T-cell lymphotropic virus (HTLV) status. The exclusion criteria for transplant is independent of eligibility for vaccination and is determined by the exclusion criteria for transplant from donors
* RECIPIENT: All subjects must have the ability to understand and the willingness to sign a written informed consent
* RECIPIENT: Participant must be willing to comply with study and/or follow-up procedures, including willingness to be followed for one year post-HCT
* RECIPIENT: Age 18 to 75 years
* RECIPIENT: Planned HCT for the treatment of the following hematologic malignancies: lymphoma (Hodgkin and non-Hodgkin), myelodysplastic syndrome, acute lymphoblastic leukemia in first or second remission, acute myeloid leukemia in first or second remission, chronic myelogenous leukemia (in first chronic or accelerated phase, or in second chronic phase), chronic lymphocytic leukemia, myeloproliferative disorders and myelofibrosis (City of Hope [COH] only). Patients with multiple myeloma are excluded
* RECIPIENT: CMV seropositive
* RECIPIENT: Planned related HCT with 8/8 (A, B, C, DRB1) high resolution HLA donor allele matching
* RECIPIENT: Conditioning and immunosuppressive regimens according to institutional guidelines are permitted
* RECIPIENT: Negative serum or urine beta-human chorionic gonadotropin (HCG) test (female patient of childbearing potential only) within two weeks of registration
* RECIPIENT: Seronegative for HIV, HCV and active HBV (surface antigen negative) within 2 months of registration
* RECIPIENT: Agreement by females of childbearing potential and males with partners of childbearing potential to use effective contraception (hormonal or barrier method or abstinence) prior to study entry and for up to 90 days post-HCT. Should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately

Exclusion Criteria:

* TRANSPLANT FROM DONOR: Unfit to undergo standard stem cell mobilization and apheresis e.g. abnormal blood counts, history of stroke, uncontrolled hypertension
* TRANSPLANT FROM DONOR: Sickling hemoglobinopathy including HbSS, HbAS, HbSC
* TRANSPLANT FROM DONOR: Positive for human immunodeficiency virus (HIV), active hepatitis B (hepatitis B virus [HBV]), hepatitis C (hepatitis C virus [HCV]) or human T-cell lymphotropic virus (HTLV-I/II). This holds true even if donors have been already vaccinated according to criteria for donor vaccination
* TRANSPLANT FROM DONOR: Donors with impaired cardiac function are excluded. Electrocardiography is routine for potential HCT donors over 60 years old and those with a history of heart disease. Subjects in whom cardiac function is abnormal (excluding 1st degree branch block, sinus brachycardia, sinus tachycardia or non-specific T wave changes) are ineligible for Triplex vaccination
* TRANSPLANT FROM DONOR: Severe psychiatric illness. Mental deficiency sufficiently severe as to make compliance with the donation procedure unlikely, and making informed consent impossible
* RECIPIENT: Any prior investigational CMV vaccine
* RECIPIENT: Experimental anti-CMV chemotherapy in the last 6 months
* RECIPIENT: Planned medications from the time of HCT to day 70 post-HCT
* RECIPIENT: Live attenuated vaccines
* RECIPIENT: Medically indicated subunit (Engerix-B for HBV; Gardasil for human papillomavirus [HPV]) or killed vaccines (e.g. influenza, pneumococcal, or allergy treatment with antigen injections)
* RECIPIENT: Allergy treatment with antigens injections
* RECIPIENT: Alemtuzumab or any equivalent in vivo T-cell depleting agent
* RECIPIENT: Antiviral medications with known therapeutic effects on CMV such as ganciclovir (GCV)/valganciclovir (VAL), FOS, Cidofovir, CMX-001, maribavir. Acyclovir has no known therapeutic efficacy against CMV and is allowable as standard of care to prevent Herpes simplex virus (HSV)
* RECIPIENT: Prophylactic therapy with CMV immunoglobulin or prophylactic antiviral CMV treatment (Letermovir is permitted). EXCEPT for low risk patients [8/8 high resolution HLA donor allele matching HCT])
* RECIPIENT: Other investigational product - concurrent enrollment in other clinical trials using any investigational new drug (IND) drugs with unknown effects on CMV or with unknown toxicity profiles is prohibited
* RECIPIENT: Other medications that might interfere with the evaluation of the investigational product
* RECIPIENT: Diagnosis with autoimmune disease
* RECIPIENT: Pregnant women and women who are lactating. The risks of CMV-MVA-Triplex to pregnant women are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother. Breastfeeding should be discontinued if the mother is enrolled on this study
* RECIPIENT: Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., social/ psychological issues, etc
* RECIPIENT: Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2022-01-22 (Actual); Study Completion 2026-07-29 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ryotaro Nakamura, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] La Rosa C, Aldoss I, Park Y, Yang D, Zhou Q, Gendzekhadze K, Kaltcheva T, Rida W, Dempsey S, Arslan S, Artz A, Ball B, Nikolaenko L, Pullarkat VA, Nakamura R, Diamond DJ. Hematopoietic stem cell donor vaccination with cytomegalovirus triplex augments frequencies of functional and durable cytomegalovirus-specific T cells in the recipient: A novel strategy to limit antiviral prophylaxis. Am J Hematol. 2023 Apr;98(4):588-597. doi: 10.1002/ajh.26824. Epub 2023 Jan 11. PMID 36594185

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Donor (Multi-peptide CMV-modified Vaccinia Ankara Vaccine) | Receipient (Multi-peptide CMV-modified Vaccinia Ankara Vaccine)
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Donor (Multi-peptide CMV-modified Vaccinia Ankara Vaccine) | Receipient (Multi-peptide CMV-modified Vaccinia Ankara Vaccine) | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [40 to 60] | 56 [44 to 60] | 53 [40 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 16
  Not Hispanic or Latino | 10 | 8 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 12 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Delayed Engraftment
Description: Time to neutrophil engraftment was defined as days from stem cell infusion to the first of three consecutive days of absolute neutrophil count ≥0.5 x 109/L. Delayed engraftment was defined as ≥20 days to neutrophil recovery.
Time Frame: Up to 1 year from stem cell infusion.
Measure: Count of Participants; unit: Participants
Groups:
- Recipients (Multi-peptide CMV-modified Vaccinia Ankara Vaccine): Participants undergo hematopoietic cell transplantation on day 0 and receive multi-peptide CMV-modified Vaccinia Ankara vaccine injection on days 28 and 56.
Arm/Group | Recipients (Multi-peptide CMV-modified Vaccinia Ankara Vaccine)
Number analyzed (Participants) | 17
Participants | 0

2. Primary Outcome: Severe (Grade III-IV) Acute Graft Versus Host Disease
Description: Acute graft versus host disease (aGvHD) happens within days or as late as 6 months after allogeneic transplants. The three main tissues that acute GVHD affects are the skin, liver, and gastrointestinal tract.
Time Frame: Up to 6 months from stem cell infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Recipients (Multi-peptide CMV-modified Vaccinia Ankara Vaccine)
Number analyzed (Participants) | 17
Participants | 2

3. Primary Outcome: Number of Recipients With Grade 3-4 Adverse Events
Description: Toxicities were assessed in recipients by Common Terminology Criteria for Adverse Events version 4.0.
Time Frame: Up to 1 year from stem cell infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | Recipients (Multi-peptide CMV-modified Vaccinia Ankara Vaccine)
Number analyzed (Participants) | 17
Participants | 0

4. Primary Outcome: Number of Donors With Grade 2-3 Adverse Events
Description: Toxicities were assessed in recipients by Common Terminology Criteria for Adverse Events version 4.0.
Time Frame: Up to 6 months after G-CSF mobilization
Measure: Count of Participants; unit: Participants
Arm/Group | Donor (Multi-peptide CMV-modified Vaccinia Ankara Vaccine)
Number analyzed (Participants) | 17
Participants | 3

5. Primary Outcome: 100-Day Non-Relapse Mortality (NRM)
Description: NRM was defined as death without recurrent or progressive disease after allogeneic transplant. Probabilities of NRM were estimated with the use of cumulative incidence curves, with relapse viewed as a competing risk.
Time Frame: From stem cell infusion up to 100 days post-HSCT (hematopoietic stem cell transplantation).
Measure: Number; unit: percentage of evaluable participants
Arm/Group | Recipients (Multi-peptide CMV-modified Vaccinia Ankara Vaccine)
Number analyzed (Participants) | 17
percentage of evaluable participants | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored/assessed from day of Triplex injection to 365 days after stem cell infusion. All-Cause Mortality was monitored/assessed up to 13 months from day of Triplex injection.
Arm/Group | Donor (Multi-peptide CMV-modified Vaccinia Ankara Vaccine) | Receipient (Multi-peptide CMV-modified Vaccinia Ankara Vaccine)
All-Cause Mortality (participants affected / at risk) | 0/17 | 2/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 2/17
Other Adverse Events (participants affected / at risk) | 16/17 | 5/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donor (Multi-peptide CMV-modified Vaccinia Ankara Vaccine) (N=17) | Receipient (Multi-peptide CMV-modified Vaccinia Ankara Vaccine) (N=17)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donor (Multi-peptide CMV-modified Vaccinia Ankara Vaccine) (N=17) | Receipient (Multi-peptide CMV-modified Vaccinia Ankara Vaccine) (N=17)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Chest pain - cardiac (Cardiac disorders) | 2 (2) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Chills (General disorders) | 3 (3) | 3 (4)
Fatigue (General disorders) | 10 (10) | 3 (3)
Fever (General disorders) | 4 (4) | 2 (2)
Hair loss (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 13 (13) | 1 (1)
Malaise (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Tenderness to Jaw area (General disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (1) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Cholesterol high (Investigations) | 0 (0) | 3 (3)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 3 (3)
White blood cell decreased (Investigations) | 0 (0) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 9 (10) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
cold (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
scalp lesions (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/52/NCT03560752/Prot_SAP_000.pdf